CLINICAL TRIAL: NCT05937334
Title: The Cohort Study for Asthma in China: an Prospective Observational Study
Brief Title: The Cohort Study for Asthma in China
Status: Recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Kewu Huang, chief physician, Beijing Chao Yang Hospital
Other Study IDs: YJXBF202201
Record Dates: First submitted 2023-04-21; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Asthma, Bronchial
MeSH Terms: conditions — Asthma | interventions — Fractional Exhaled Nitric Oxide Testing; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood sample, Induced sputum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: lung function test, chest CT, induced sputum, blood routine test, IgE test, FeNO test, six minutes walk test, questionnaires for asthma — lung function test, chest CT, induced sputum, blood routine test, IgE test, FeNO test, six minutes walk test, questionnaires for asthma were performed. All interventions was made according to routine diagnosis and treatment.

SUMMARY:
The study is to establish a standardized asthma cohort study, build an information network platform system and a biospecimen bank for asthma cohort, establish clear follow-up standards and norms, observe the asthma outcomes and identify biomarkers to predict asthma outcomes.

DETAILED DESCRIPTION:
This is a single center observational prospective longitudinal cohort study to establish a standardized asthma cohort, consisting of 400 patients with asthma. Baseline data including lung function test, chest CT, induced sputum, etc. was collected and the patients were followed up for 2 or more years. Subjects who met the 2023 GINA diagnostic criteria for asthma and were able to participate in the study according to the protocol and sign the informed consent were included. No additional investigational drugs will be applied to the patients. Blood samples are transported to designated laboratories for safekeeping and biomarker testing. We aimed to explore the mechanism of biomarkers involved in asthma pathogenesis and identify treatable traits related to disease outcome. Full analysis set will be used for all analyses. Missing data will be analyzed as it is. Statistical analysis will be conducted by epidemiology & statistics work group from Chinese Academy of Sciences, using SAS and SUDAAN software. An electronic data capture system will be used in this study. Paper-based questionnaire administration will also be used. Questionnaire variables will be checked before data entry. During the study, PI will be in charge of the monitoring of the whole procedure. Working group will do the data cleaning and data analyzing.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Meet the 2023 edition of GINA asthma diagnostic criteria
* Subjects must sign informed consent prior to study participation, participate in the study according to the protocol and follow up for 2 years

Exclusion Criteria:

* Suffering from other massive lung tissue destructive diseases such as severe bronchiectasis and tuberculosis
* Severe pleural disease and/or sternal and rib lesions
* Serious uncontrolled disease of other system
* Thoracic or abdominal surgery in the past 3 months
* Eye surgery in the past three months
* Retina detachment
* Myocardial infarction within the last 3 months
* Hospitalized for heart disease within the past 3 months
* Ongoing anti-tuberculosis treatment
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 400 subjects will be recruited from Beijing Chao-Yang Hospital, Capital Medical University. They are over 18 years old, meet the 2023 version of GINA asthma diagnostic criteria, can participate in the study according to the protocol, and sign informed consent before participating in the study.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test(ACT) | 2 years
  As)thma control was assessed by Asthma Control Test(ACT)
Asthma Control Questionnaire(ACQ) | 2 years
  sthma control was assessed by Asthma Control Questionnaire(ACQ)
Induced sputum analysis | 2 years
  Identification of asthma endotypes was based on Induced sputum analysis

SECONDARY OUTCOMES:
Prognosis prediction of asthma with specific treatment regimen | 2 years
  Prognosis prediction of asthma with specific treatment regimen was based on different phenotypes and biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Kewu Huang, M.D., Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverstein NJ, Huh JR. Interleukin-17: Why the Worms Squirm. Immunity. 2017 Mar 21;46(3):347-349. doi: 10.1016/j.immuni.2017.03.007. PMID 28329701
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Huang K, Yang T, Xu J, Yang L, Zhao J, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Chen Y, Sun T, Shan G, Lin Y, Xu G, Wu S, Wang C, Wang R, Shi Z, Xu Y, Ye X, Song Y, Wang Q, Zhou Y, Li W, Ding L, Wan C, Yao W, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Wang Z, Chen Z, Bu X, Zhang H, Zhang X, An L, Zhang S, Zhu J, Cao Z, Zhan Q, Yang Y, Liang L, Tong X, Dai H, Cao B, Wu T, Chung KF, He J, Wang C; China Pulmonary Health (CPH) Study Group. Prevalence, risk factors, and management of asthma in China: a national cross-sectional study. Lancet. 2019 Aug 3;394(10196):407-418. doi: 10.1016/S0140-6736(19)31147-X. Epub 2019 Jun 20. PMID 31230828
- [Background] Baptist AP, Busse PJ. Asthma Over the Age of 65: All's Well That Ends Well. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):764-773. doi: 10.1016/j.jaip.2018.02.007. PMID 29747982
- [Background] Lange P, Colak Y, Ingebrigtsen TS, Vestbo J, Marott JL. Long-term prognosis of asthma, chronic obstructive pulmonary disease, and asthma-chronic obstructive pulmonary disease overlap in the Copenhagen City Heart study: a prospective population-based analysis. Lancet Respir Med. 2016 Jun;4(6):454-62. doi: 10.1016/S2213-2600(16)00098-9. Epub 2016 Apr 6. PMID 27061878
- [Background] Fingleton J, Huang K, Weatherall M, Guo Y, Ivanov S, Bruijnzeel P, Zhang H, Wang W, Beasley R, Wang C; NZ-China Study Group. Phenotypes of symptomatic airways disease in China and New Zealand. Eur Respir J. 2017 Dec 7;50(6):1700957. doi: 10.1183/13993003.00957-2017. Print 2017 Dec. PMID 29217598
- [Background] Bai TR, Vonk JM, Postma DS, Boezen HM. Severe exacerbations predict excess lung function decline in asthma. Eur Respir J. 2007 Sep;30(3):452-6. doi: 10.1183/09031936.00165106. Epub 2007 May 30. PMID 17537763
- [Background] Vale-Pereira S, Todo-Bom A, Geraldes L, Schmidt-Weber C, Akdis CA, Mota-Pinto A. FoxP3, GATA-3 and T-bet expression in elderly asthma. Clin Exp Allergy. 2011 Apr;41(4):490-6. doi: 10.1111/j.1365-2222.2010.03640.x. Epub 2010 Nov 28. PMID 21114556
- [Background] Dunn RM, Busse PJ, Wechsler ME. Asthma in the elderly and late-onset adult asthma. Allergy. 2018 Feb;73(2):284-294. doi: 10.1111/all.13258. Epub 2017 Sep 7. PMID 28722758

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT05937334/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT05937334/ICF_001.pdf